CLINICAL TRIAL: NCT01646086
Title: Weight Tracking and Weight Loss Outcomes: Establishing the Standard of Care
Acronym: Tracking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1106S01462; 1R01DK093586 (NIH)
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Weight Loss
Keywords: Weight Loss; Self-Weighing; Weight Tracking
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- weekly weight tracking (Experimental): 12 month behavioral weight loss intervention
  Interventions: Behavioral: 12 month behavioral weight loss intervention
- daily weight tracking (Active Comparator): 12 month behavioral weight loss intervention
  Interventions: Behavioral: 12 month behavioral weight loss intervention
- no weight tracking (Active Comparator): 12 month behavioral weight loss intervention
  Interventions: Behavioral: 12 month behavioral weight loss intervention

INTERVENTIONS:
Behavioral: 12 month behavioral weight loss intervention — The intervention for all groups will follow a standard behavioral weight loss protocol. Participants will meet in groups of up to 20 persons; groups will meet weekly for the first six months, then biweekly for two months and monthly for the remaining four months of the 12-month treatment period. Session content will be centered on behavioral goal setting and attention to caloric intake and physical activity. Participants will be asked to keep daily diet and physical activity logs.

SUMMARY:
To achieve the long term goal of strengthening behavioral weight loss programs, the purpose of this project is to test an enhanced, daily weight tracking instruction against the current standard of care (weekly weight tracking) and an alternative mode of care (no weight tracking).

The investigators postulate that daily weight tracking will boost ongoing awareness of and engagement in dietary intake and physical activity monitoring, thus improving weight loss outcomes. The central hypothesis of the study is that daily weight tracking will improve weight loss processes and outcomes relative to less frequent weight tracking, without adverse effects.

DETAILED DESCRIPTION:
Given the pernicious reach of obesity and the evidence that current behavioral treatments are modestly effective at changing weight, efforts to refine behavioral recommendations in order to improve weight loss interventions are crucial. Frequency of tracking body weight presents itself as a prime target for behavioral enhancement during weight loss. Daily self-monitoring (e.g., of dietary intake and physical activity) is already well-established as a central component of the behavioral weight loss process. However, the current standard of care in behavioral weight loss with regard to weighing is weekly tracking of weight, and some programs caution against any weight tracking. It has been suggested that frequent weight tracking may have a negative impact on mental health and outcomes during weight loss, but there are minimal data that address this concern experimentally in the context of an active weight loss program. Observational evidence from behavioral weight control trials and community studies suggests that greater frequency of tracking weight is associated with better weight outcomes. Stronger experimental evidence is needed to establish a causal link between weight tracking and weight outcomes and to elucidate the impact on mental health during weight loss. To achieve the long-term goal of strengthening behavioral weight loss programs, the purpose of this project is to test an enhanced, daily weight tracking instruction against the current standard of care (weekly weight tracking) and an alternate model of care with very limited data (no weight tracking). In pursuit of study goals, 336 overweight and obese adults will be recruited and randomized to one of three 12-month weight loss interventions with a 12-month follow-up (24 months total time in study): the standard of care (weekly weight tracking during weight loss), an enhanced condition (daily weight tracking during weight loss), or a comparison condition (no weight tracking during weight loss). The rationale behind this proposal is that within the context of social ecology and a social-cognitive framework of behavior change, enhancement of this key environmental feature (i.e., the weight tracking environment) during weight loss will contribute to success by promoting self-efficacy for this critical behavior. Specific aims of the study will seek to determine the effects of weight tracking frequency on the weight loss process and outcomes, as well as to elucidate the effects of weight tracking frequency on mental health during weight loss. This study will have the expected outcome of enhancing the standard of care for weight loss, leading to better weight control for overweight and obese adults and thus directly mitigating the public health impact of the obesity crisis.

ELIGIBILITY:
Inclusion Criteria:

* women and men
* 18-64 years of age
* BMI between 25.0 and 39.9 kg/m2 (overweight to obese)
* interest in joining a weight loss program
* have a computer, email, and wifi connection at home
* live in the Minneapolis/Saint Paul, Minnesota area

Exclusion Criteria:

* weight in the underweight to low normal (BMI < 22) or morbidly obese (BMI > 35) ranges
* current eating disorder or history of eating disorders
* current major depression or psychotic disorder diagnosis
* current cardiovascular disease or diabetes diagnosis
* current participation in a weight loss program
* current pregnancy
* previous weight loss surgery

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 339 (Actual)
Dates: Start 2012-07; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight Over Time | baseline, 6 months, 12 months, 18 months, and 24 months
  Weight (in kilograms) will be measured by study staff using a calibrated digital scales with participants wearing light clothing and no shoes. Height (in centimeters) will be measured by study staff at baseline only using a portable stadiometer. BMI (kg/m2) will be calculated from these measurements

SECONDARY OUTCOMES:
Demographic Measures | baseline
  Age, sex, marital status, employment status, income level (categorical), race, and ethnicity will be assessed by self-report at baseline
Weight Tracking and Self-Monitoring Adherence | throughout intervention
  Self-monitoring data on diet, physical activity, and weight from electronic or paper records will be recorded by interventionists at each session by compiling printouts of electronic records from websites supported by electronic monitoring tools, and by photocopying paper diaries for participants without electronic monitoring tools.
Perceptions of Weight Tracking | 6 months, 12 months, 18 months, and 24 months
  Participants complete an 8-item questionnaire to assess beliefs about their weight tracking assignment during the study. The measure asks participants to rate daily, weekly, or no weight tracking in terms of ease, interest level, ability to remember, awareness, reward value, usefulness, understanding, and how motivated they are to engage in their assigned weight tracking frequency. These items measure aspects of cue strength and motivational value, both of which are important to the process of behavior modification within a social-ecological frame (DiClemente et al., 2001; Elder et al., 2007)
Barriers to Weight Tracking | baseline, 6 months, 12 months, 18 months, and 24 months
  To elucidate factors that may impede engagement in daily or weekly weight tracking, participants will complete an assessment of perceived barriers to tracking weight. Items for this measure were adapted from a measure of barriers to diet and exercise developed by a member of the research team and used in numerous weight loss studies These items will provide feedback on factors that may interfere with weight tracking and will provide guidance for adaptation and use of weight tracking instructions for future interventions.
Self-Efficacy for Weight Loss Behaviors | baseline, 6 months, 12 months, 18 months, and 24 months
  Self-efficacy for dietary intake, physical activity, and weight tracking behaviors will be assessed using a 15-item scale developed by members of the research team (Linde et al., 2006).
Routine Health Habits | baseline, 12 months, and 24 months
  Participants will complete brief screening items developed for the study to assess smoking status, sedentary behavior (television viewing) and days per week of engaging in weight control behaviors, including diet and physical activity monitoring. Weight tracking frequency (never, every other month, monthly, weekly, or daily) and number of body weight scales at home will also be assessed.
Dietary Intake | baseline, 6 months, 12 months, 18 months, and 24 months
  The Diet History Questionnaire (DHQ, 2010) is a food frequency questionnaire (FFQ) that assesses usual intake and portion size of 124 foods. Responses are scored and analyzed using proprietary Diet*Calc software, which provides reasonable and valid estimates of macronutrient and caloric intake compared to 24-hour recall administrations (Millen et al., 2006) and alternate FFQ protocols (Subar et al., 2001). A subset of 168 participants (50%; 56 per treatment condition) will be randomized at baseline to a 24-hr dietary recall protocol.
Physical Activity | baseline, 6 months, 12 months, 18 months, and 24 months
  The Paffenbarger Activity Questionnaire (PAQ; Paffenbarger et al., 1978) will be administered to provide an estimate of calories expended per week in leisure time physical activities. The PAQ has been associated with weight loss outcomes in intervention trials (e.g., Harris et al., 1994). A subset of 168 participants (50%; 56 per treatment condition) will be randomized to a 7-day accelerometer protocol at baseline and 12 months to enhance physical activity measurement during active weight loss, to elucidate any changes in daily patterning of activity that might occur during intervention.
Body Image | baseline, 6 months, 12 months, 18 months, and 24 months
  The Appearance Evaluation subscale of the Multidimensional Body-Self-Relations Questionnaire will assess body image.
Self-Esteem | baseline, 6 months, 12 months, 18 months, and 24 months
  The Rosenberg Self-Esteem Scale (Rosenberg, 1979) will rate global self-esteem and will be used to track well-being during the study.
Depression | baseline, 6 months, 12 months, 18 months, and 24 months
  The Beck Depression Inventory (BDI-II) will assess depressive symptoms that may change over the course of the study period.
Anxiety | baseline, 6 months, 12 months, 18 months, and 24 months
  The Beck Anxiety Inventory (BAI) will assess anxiety symptoms that may change over the study.
Mood States | baseline, 6 months, 12 months, 18 months, and 24 months
  The Positive and Negative Affect Schedule - Expanded Form (PANAS-X) will be administered as a momentary assessment of mood during randomly selected intervention sessions. The measure, consisting of 60 adjectives that are rated on a five-point Likert scale (from 1=very slightly or not at all to 5=extremely), assesses positive and negative affect, basic negative emotions (fear, hostility, guilt, sadness), basic positive emotions (joviality, self-assurance, attentiveness), and additional mood states (shyness, fatigue, serenity, surprise).
Life Events | baseline, 12 months, and 24 months
  The Life Experiences Survey (Sarason et al., 1978) will assess a broad range of life changes and events that could affect participation in weight tracking or other study recommendations. We expect that participants who endorse a greater number of stressful life events will have poorer adherence, will be less able to maintain tracking diaries, and will experience greater negative affect relative to those with fewer life events during the study (Dunkley et al., 2003; Sarason et al., 1978).
Eating Disorder Symptoms | baseline, 6 months, 12 months, 18 months, and 24 months
  Measures used to screen participants prior to study entry will be repeated during the trial for ongoing monitoring. These include the Questionnaire on Eating and Weight Patterns to assess binge eating, and the SCOFF Eating Disorder Screening Questionnaire to assess presence of symptoms associated with anorexia or bulimia.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Linde, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Crane MM, Gavin K, Wolfson J, Linde JA. How Accurate are Recalls of Self-Weighing Frequency? Data from a 24-Month Randomized Trial. Obesity (Silver Spring). 2018 Aug;26(8):1296-1302. doi: 10.1002/oby.22239. Epub 2018 Aug 1. PMID 30070045
- See also: Click here for more information about eligibility criteria — http://www.epi.umn.edu/tracking/